CLINICAL TRIAL: NCT03063658
Title: Comparison of the Postoperative Analgesia Effectiveness of Preemptive Intravenous Ibuprofen and Paracetamol in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Comparison of the Effectiveness of Preemptive Paracetamol and Ibuprofen in Acute Postoperative Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Menekse Ozcelik, M.D, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16-827-16
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Acute Pain; Postoperative Pain
Keywords: Ibuprofen; Paracetamol; Laparoscopic cholecystectomy; Morphine; Visual analog scale
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paracetamol (Active Comparator): Paracetamol (Paracerol) 1 gram will be administered intravenously. The first dose will be infused for 10 minutes after the induction of anesthesia and before the first surgical incision. The remaining three doses will be administered every 6 hours for postoperative 24 hours.
  Interventions: Drug: Paracetamol
- Ibuprofen (Active Comparator): Ibuprofen (Intrafen) 800 mg will be administered intravenously. The first dose will be infused for 10 minutes after the induction of anesthesia and before the first surgical incision. The remaining three doses will be administered every 6 hours for postoperative 24 hours.
  Interventions: Drug: Ibuprofen 800 mg

INTERVENTIONS:
Drug: Paracetamol — The first dose of 1 gr intravenous paracetamol will be administered preoperatively and the remaining three doses will be given each six hours in the early postoperative period.
  Arms: Paracetamol
Drug: Ibuprofen 800 mg — The first dose of 800 mg intravenous ibuprofen will be administered preoperatively and the remaining three doses will be given each six hours in the early postoperative period.
  Arms: Ibuprofen

SUMMARY:
This study will evaluate two different analgesic regimen used for acute postoperative pain.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is a type of surgery that causes moderate postoperative pain. Paracetamol and non-steroid anti-inflammatory analgesics plus opioids are the mainstay treatment options of the moderate postoperative pain. These drugs are the most common used analgesics to ameliorate this type of pain and to reduce the consumption of opioids and their side effects.

Ibuprofen is a well-known anti-inflammatory drug and has been used as an oral formula for a long time. Few studies using its new intravenous formula had been conducted to evaluate its effectiveness for mixed type of surgeries . However, its intravenous formula has not been studied for laparoscopic cholecystectomy. Therefore, this study will compare the effects of postoperative analgesic potencies of preemptive intravenous paracetamol and ibuprofen in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologist Functional Status 1-2
2. Body mass index smaller than 30
3. Undergoing laparoscopic cholecystectomy
4. Age between 18-60 years

Exclusion Criteria:

1. Age under 18, above 60
2. Weight under 40 kg
3. Body mass index above 30
4. Contraindication for opioid and non-steroid anti-inflammatory drug usage
5. Allergy against paracetamol, opioids and anti-inflammatory drugs
6. Peptic ulcer
7. Tendency to bleeding
8. Pregnancy or breast feeding
9. Moderate or severe renal, hepatic or cardiac insufficiency
10. Coronary artery disease
11. Asthma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | The first 24 hours after the completion of the surgery
  Total morphine consumption during the 24 hours of early postoperative period

SECONDARY OUTCOMES:
VAS scores | The first 24 hours after the completion of the surgery
  VAS scores at rest, at movement, at cough will be evaluated during the first 24 hours of early postoperative period
Morphine side effects | The first 24 hours after the completion of the surgery
  Morphine side effects such as nausea, vomiting, pruritus, constipation, urinary retention will be evaluated during the first 24 hours of early postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Zekeriyya Alanoglu, Professor, Principal Investigator — Ankara University Department of Anesthesiology and Intensive Care Medicine
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara University Faculty of Medicine, Ankara
  - Ankara University School of Medicine, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singla N, Rock A, Pavliv L. A multi-center, randomized, double-blind placebo-controlled trial of intravenous-ibuprofen (IV-ibuprofen) for treatment of pain in post-operative orthopedic adult patients. Pain Med. 2010 Aug;11(8):1284-93. doi: 10.1111/j.1526-4637.2010.00896.x. Epub 2010 Jun 30. PMID 20609131
- [Background] Gago Martinez A, Escontrela Rodriguez B, Planas Roca A, Martinez Ruiz A. Intravenous Ibuprofen for Treatment of Post-Operative Pain: A Multicenter, Double Blind, Placebo-Controlled, Randomized Clinical Trial. PLoS One. 2016 May 6;11(5):e0154004. doi: 10.1371/journal.pone.0154004. eCollection 2016. PMID 27152748
- [Background] Gan TJ, Candiotti K, Turan A, Buvanendran A, Philip BK, Viscusi ER, Soghomonyan S, Bergese SD; Intravenous Ibuprofen Surgical Surveillance Trial Investigational Sites. The shortened infusion time of intravenous ibuprofen, part 2: a multicenter, open-label, surgical surveillance trial to evaluate safety. Clin Ther. 2015 Feb 1;37(2):368-75. doi: 10.1016/j.clinthera.2014.12.006. Epub 2015 Jan 13. PMID 25592331